CLINICAL TRIAL: NCT07066189
Title: Lifestyle, Exercise, And Nutrition (LEAN) Trial on Pathologic Complete Response in Triple Negative Breast Cancer (TNBC)
Brief Title: Lifestyle, Exercise, And Nutrition (LEAN) Trial on Pathologic Complete Response in TNBC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: Breast Cancer Research Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2000039695
Record Dates: First submitted 2025-06-24; First posted 2025-07-15 (Actual); Last update posted 2025-10-29 (Actual); Status verified 2025-10

CONDITIONS: Triple Negative Breast Cancer
Keywords: Exercise; Diet; Pathologic complete response; Neoadjuvant therapy
MeSH Terms: conditions — Triple Negative Breast Neoplasms; Motor Activity; Pathologic Complete Response | interventions — Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The following study personnel will be masked to participant study arm: the staff performing DXA scan and blood processing/biomarker evaluation. The staff performing clinic measures, study staff reviewing forms and entering data, the PI and Co-Is, the statistician, study manager, and interventionists will be unblinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise and Medical Nutrition (Experimental): Women randomized to the intervention will receive 10, 30-minute sessions spread out over the course of their neoadjuvant therapy and in the weeks leading up to surgery. In weeks in which one of the 10 counseling sessions is not scheduled the interventionist will observe the participant in an exercise session via zoom, or check in with the participant by phone regarding their exercise. The intervention will continue until the day prior to the last chemotherapy infusion.
  Interventions: Behavioral: Exercise and Medical Nutrition
- Usual care (No Intervention): Contact limited to study assessments.

INTERVENTIONS:
Behavioral: Exercise and Medical Nutrition — 10, 30-minute sessions spread out over the course of their neoadjuvant therapy and in the weeks leading up to surgery. On weeks counseling is not scheduled an exercise session will be observed.
  Arms: Exercise and Medical Nutrition

SUMMARY:
The purpose of this study is to examine whether a nutrition and exercise program can improve pathologic complete response (pCR) in women with triple-negative breast cancer (TNBC) receiving chemo-immunotherapy before surgery. Pathologic complete (pCR) response means that no cancer in the breast is seen after chemotherapy.

DETAILED DESCRIPTION:
Women with stage II-III triple-negative breast cancer (TNBC) undergoing neoadjuvant chemo-immunotherapy will be enrolled in the study. Following screening, consent, and baseline assessment, participants will be randomized to either the intervention group (nutrition and exercise counseling) or the usual care group. Participants randomized to the intervention group will complete weekly remote sessions with the interventionist throughout the duration of chemotherapy. Each counseling session will last about 30 minutes and will be conducted remotely. The exercise regimen is home-based.

Study activities include completing surveys and attending two in-person study visits, each of which will include a blood draw, a 6-minute walk test to assess aerobic capacity and endurance, and a Dual Energy X-Ray Absorptiometry (DXA) scan to measure body composition.

The primary outcome is the pathologic complete response.

Researchers will also compare the exercise and nutrition program to usual care to determine if the program improves residual cancer burden, symptoms related to cancer treatment, body composition, and blood biomarkers.

ELIGIBILITY:
Inclusion Criteria:

1. Female aged 18 years or older.
2. Have a diagnosis of stage II or III Triple Negative Breast Cancer (TNBC).
3. Be scheduled to receive neoadjuvant chemo-immunotherapy.
4. Be physically able to walk.
5. Be able to complete forms, understand instructions and read in English.
6. Agree to be randomly assigned to either group.
7. Have clearance from oncologist to participate.
8. Not exercising (less than 150 min/week).
9. Not consuming more than 7 fruits and vegetable/week.

Exclusion Criteria:

1. Having already started a 2nd chemotherapy cycle.
2. Pregnancy or intention to become pregnant.
3. Presence of dementia or major psychiatric disease.
4. Recent (past year) stroke, myocardial infarction, or congestive heart failure.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2025-10-17 (Actual); Primary Completion 2029-10 (Estimated); Study Completion 2029-10 (Estimated)

PRIMARY OUTCOMES:
Pathologic Complete Response (pCR) | Post breast cancer surgery, an average of 6 months
  Pathologic Complete Response (pCR) is defined as having no invasive residual disease in the breast or regional lymph nodes after completing neoadjuvant chemotherapy (ypT0 ypN0 or ypT0/is ypN0)

SECONDARY OUTCOMES:
Residual Cancer Burden (RCB) | Post breast cancer surgery, an average of 6 months
  Residual Cancer Burden (RCB) is a continuous pCR measure.

OTHER OUTCOMES:
Healthy Eating Index (HEI) | Baseline to end of first line chemotherapy, on average 6 months
  Healthy Eating Index (HEI) will be will be estimated using the self-reported food frequency questionnaire developed by Fred Hutchinson Cancer Center.
Physical activity | Baseline to end of first line chemotherapy, on average 6 months
  Self-reported minutes per week of moderate- to vigorous-intensity physical activity will be estimated using the modifiable physical activity questionnaire.
Patient reported toxicities | Baseline to end of first line chemotherapy, on average 6 months
  Participants will be asked to complete the Patient-Reported Outcomes version of the Common Terminology Criteria for Adverse Events (PRO-CTCAE) survey at baseline, 2-months, 4-months and the end of chemotherapy.
Physical function | Baseline to end of first line chemotherapy, on average 6 months
  Participants will be asked to complete the Patient-Reported Outcomes Measurement Information System (PROMIS)-29 survey.
Fatigue | Baseline to end of first line chemotherapy, on average 6 months
  Participants will be asked to complete the Patient-Reported Outcomes Measurement Information System (PROMIS)-29 survey.
Neuropathy | Baseline to end of first line chemotherapy, on average 6 months
  Participants will be asked to complete the Functional Assessment of Cancer Therapy (FACT)-neuropathy subscale (FACT-Ntx).
Malnutrition | Baseline to end of first line chemotherapy, on average 6 months
  Participants will be asked to complete the Patient-Generated Subjective Global Assessment (PG-SGA).
Aerobic capacity | Baseline to end of first line chemotherapy, on average 6 months
  Participants will be asked to complete a 6-minute walk test.
Lean mass | Baseline to end of first line chemotherapy, on average 6 months
  Participants will be asked to complete a Dual Energy X-Ray Absorptiometry (DXA) scan
Percent fat | Baseline to end of first line chemotherapy, on average 6 months
  Participants will be asked to complete a Dual Energy X-Ray Absorptiometry (DXA) scan

CONTACTS AND LOCATIONS:
Overall Officials: Melinda Irwin, Principal Investigator — Yale University
Locations (1):
- Yale University, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No